CLINICAL TRIAL: NCT00667173
Title: A Phase 2, Multi-Center, Evaluator-Blind, Randomized, Vehicle-Controlled Clinical Study to Assess the Safety and Efficacy of IDP-115 in the Treatment of Rosacea
Brief Title: A Clinical Study Evaluating the Safety and Efficacy of IDP-115 in Patients With Rosacea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPSI-IDP-115-P2-01
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: IDP-115
- 2 (Placebo Comparator)
  Interventions: Drug: Vehicle
- 3 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: IDP-115 — Topical application for 12 weeks
  Arms: 1
Drug: Vehicle — Topical application for 12 weeks
  Arms: 2
Drug: Vehicle — Topical application for 12 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of IDP-115 in treating patients with rosacea.

ELIGIBILITY:
Inclusion Criteria:

* Presence of facial rosacea
* Presence of inflammatory lesions

Exclusion Criteria:

* Dermatological conditions of the face that could interfere with clinical evaluations
* Known history of photosensitivity disorders (such as lupus erythematosus or polymorphous light eruption)
* Female subjects who are pregnant, nursing, planning a pregnancy, or become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the number of inflammatory lesions | 12 weeks
Improvement from baseline in global severity | 12 weeks

SECONDARY OUTCOMES:
Change from baseline in erythema | 12 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Therapeutics Clinical Research, San Diego, California
  - Solano Clinical Research, Vallejo, California
  - Cherry Creek Dermatology Research Inc., Denver, Colorado
  - FXM Research Corp., Miami, Florida
  - MedaPhase Inc., Newnan, Georgia
  - Henry Ford Medical Center, Detroit, Michigan
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - University Dermatology Consultants, Inc., Cincinnati, Ohio
  - DermResearch, Inc., Austin, Texas